CLINICAL TRIAL: NCT02021890
Title: A Standard Ballroom and Latin Dance Program to Improve Fitness and Adherence to Physical Activity in Individuals With Type 2 Diabetes and Obesity
Brief Title: Efficacy Study of Standard Ballroom and Latin Dance Program in Type 2 Diabetes and Obesity
Acronym: BALLANDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: General Hospital, Gavardo (Unknown); Villa Garda Hospital (Other)
Responsible Party: Principal Investigator, Giulio Marchesini R., M.D., Professor of Dietetics, University of Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BALLANDO
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes; Obesity
Keywords: Dance; Physical activity; Physical fitness; Weight loss
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Motor Activity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ballroom and Latin dance program (Experimental): two-hour dancing session twice a week
  Interventions: Behavioral: Dance program
- Self-selected physical activity (Active Comparator): self-selected program of physical activity
  Interventions: Behavioral: Self-selected physical activity

INTERVENTIONS:
Behavioral: Dance program — two-hour dancing session twice a week, led by instructors in a private hall of a disco. Both solo and partner and group dances were performed during each session: an initial one-hour activity, chaired by two instructors who taught new steps and choreographies to patients (both individually and in group), was followed by a second hour, when patients danced in pairs both Latin and standard ballroom music
  Arms: ballroom and Latin dance program
Behavioral: Self-selected physical activity — gym sessions (with the support of sports associations), exercising at home (cycling, stepping) or walking, jogging or cycling outside with/without group support
  Arms: Self-selected physical activity

SUMMARY:
to test the metabolic and clinical effects of a 6-month program of dancing in subjects with type 2 diabetes and/or obesity, chronically cared for in two diabetes/metabolic units. Self-selection of the leisure time activity program was allowed to increase adherence to the physical activity programs.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes in fairly good metabolic control (glycosylated hemoglobin (HbA1c) < 8.5%) and/or obesity (Body Mass Index (BMI) ≥ 30 kg/m2 or waist circumference >94 cm in males, >80 in females), with/without prediabetes or minor alterations of HbA1c.

Exclusion Criteria:

* previous cardiovascular events, muscle-skeletal problems reducing physical ability, any general condition limiting systematic adherence

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
5% reduction in BMI or waist circumference | 3 months
5% reduction in BMI or waist circumference | 6 months
improved physical fitness (physical activity exceeding 10 MET-hour/week | 3 months
improved physical fitness (physical activity exceeding 10 MET-hour/week | 6 months

SECONDARY OUTCOMES:
0.3% reduction of HbA1c in the presence of diabetes | 3 months
0.3% reduction of HbA1c in the presence of diabetes | 6 months
10% increase in 6-min walk test | 3 months
10% increase in 6-min walk test | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Unit of Metabolic Diseases and Clinical Dietetics, "Alma Mater Studiorum" University, Bologna, Bologna
  - Unit of Endocrinology and Diabetology, General Hospital, Gavardo, Brescia

REFERENCES:
- [Derived] Mangeri F, Montesi L, Forlani G, Dalle Grave R, Marchesini G. A standard ballroom and Latin dance program to improve fitness and adherence to physical activity in individuals with type 2 diabetes and in obesity. Diabetol Metab Syndr. 2014 Jun 22;6:74. doi: 10.1186/1758-5996-6-74. eCollection 2014. PMID 25045404